CLINICAL TRIAL: NCT02687503
Title: Impact of Probiotic Use on Immune Cell Function in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0884; A536700 (Other: UW Madison); SMPH\PEDIATRICS\PEDIATRICS (Other: UW Madison)
Record Dates: First submitted 2016-01-25; First posted 2016-02-22 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-03

CONDITIONS: Respiratory Tract Infections
Keywords: Immune system; Probiotics
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daily dose of probiotic (Other): All children enrolled into the study will receive a daily dose of probiotic
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — All children will receive a daily dose of probiotic (10⁹ cfu of L.acidophilus NCFM and B. lactis, Bi-07), a commercially available probiotic. Parents will give probiotic in 1 ounce of milk or water once a day for 30 days in an open label fashion.

SUMMARY:
Probiotics are microorganisms that are believed to provide health benefits when consumed. The term probiotic is currently used to name ingested microorganisms associated with beneficial effects to humans and animals. Probiotics are popularized in the lay literature for many different clinical problems. They have been studied in infants and children as a preventive or treatment for a variety of infections. Studies on the medical benefits of probiotics have yet to reveal a cause-effect relationship, and their medical effectiveness has yet to be conclusively proven for most of the studies conducted thus far. The putative benefit of probiotics in the prevention of infection relates to potential benefits to the innate and adaptive immune systems of infants.

The goals of this investigation are to study immune system cell function and microbiome in children who are taking probiotics.

To accomplish this goal, we propose a pilot study for which we will obtain blood and nasopharyngeal and stool samples prior to and post probiotic use in children greater than 12 months-36 months over a 27-38 day period

ELIGIBILITY:
Inclusion Criteria

* Healthy children greater than 12 months-36 months of age
* English speaking parent
* Child has not received a live vaccine such as MMR or Varicella in the past 2 weeks

Exclusion Criteria

* Asthma/allergic rhinitis
* Premature birth (< 36 weeks gestation)
* Known to be lactose intolerant
* Immunodeficiency or any underlying problem requiring the use of steroids or other immunosuppressive agents
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) such as ibuprofen in the last 2 weeks
* Currently taking probiotics, have received probiotics in the previous two weeks or are unwilling to refrain from the use of non-study probiotics during the next 30 days
* Any antibiotic treatment in the last 2 weeks
* Conditions which might interfere with dispersion of the probiotic after oral administration such as short gut or anomalies of the digestive tract
* Concurrently participating in another clinical study, in which the child has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Innate immune cell multiparameter flow cytometry assay | 3 months
  The primary measurement will be plasmacytoid dendritic cell responses to various TLR agonists (CpGA, R848) and intact human rhinovirus. Variables measured will include pDC frequency, frequency of IFN-alpha and TNF-alpha producing cells and geometric mean fluorescence intensity of these cytokines using an optimized and standardized multi-parameter flow cytometry assay.

SECONDARY OUTCOMES:
Isolation of peripheral blood mononuclear cells (PBMC) by density gradient | 3 months
  Multi-parameter flow cytometry will be used to determine the frequency of CD25+CD127-/loFoxp3+CD4+ T cells. Function will be indirectly CD25+ determined by quantifying the level of TSDR demethylation in Treg cells.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UW Health 20 S. Park Clinic, Madison, Wisconsin
  - UW Health West Towne Clinic, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olenec JP, Kim WK, Lee WM, Vang F, Pappas TE, Salazar LE, Evans MD, Bork J, Roberg K, Lemanske RF Jr, Gern JE. Weekly monitoring of children with asthma for infections and illness during common cold seasons. J Allergy Clin Immunol. 2010 May;125(5):1001-1006.e1. doi: 10.1016/j.jaci.2010.01.059. Epub 2010 Apr 14. PMID 20392488
- [Background] Hatakka K, Savilahti E, Ponka A, Meurman JH, Poussa T, Nase L, Saxelin M, Korpela R. Effect of long term consumption of probiotic milk on infections in children attending day care centres: double blind, randomised trial. BMJ. 2001 Jun 2;322(7298):1327. doi: 10.1136/bmj.322.7298.1327. PMID 11387176
- [Background] Hojsak I, Abdovic S, Szajewska H, Milosevic M, Krznaric Z, Kolacek S. Lactobacillus GG in the prevention of nosocomial gastrointestinal and respiratory tract infections. Pediatrics. 2010 May;125(5):e1171-7. doi: 10.1542/peds.2009-2568. Epub 2010 Apr 19. PMID 20403940
- [Background] Lin JS, Chiu YH, Lin NT, Chu CH, Huang KC, Liao KW, Peng KC. Different effects of probiotic species/strains on infections in preschool children: A double-blind, randomized, controlled study. Vaccine. 2009 Feb 11;27(7):1073-9. doi: 10.1016/j.vaccine.2008.11.114. Epub 2008 Dec 27. PMID 19114073
- [Background] Maldonado J, Canabate F, Sempere L, Vela F, Sanchez AR, Narbona E, Lopez-Huertas E, Geerlings A, Valero AD, Olivares M, Lara-Villoslada F. Human milk probiotic Lactobacillus fermentum CECT5716 reduces the incidence of gastrointestinal and upper respiratory tract infections in infants. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):55-61. doi: 10.1097/MPG.0b013e3182333f18. PMID 21873895
- [Background] Merenstein D, Murphy M, Fokar A, Hernandez RK, Park H, Nsouli H, Sanders ME, Davis BA, Niborski V, Tondu F, Shara NM. Use of a fermented dairy probiotic drink containing Lactobacillus casei (DN-114 001) to decrease the rate of illness in kids: the DRINK study. A patient-oriented, double-blind, cluster-randomized, placebo-controlled, clinical trial. Eur J Clin Nutr. 2010 Jul;64(7):669-77. doi: 10.1038/ejcn.2010.65. Epub 2010 May 19. PMID 20485304
- [Background] Taipale T, Pienihakkinen K, Isolauri E, Larsen C, Brockmann E, Alanen P, Jokela J, Soderling E. Bifidobacterium animalis subsp. lactis BB-12 in reducing the risk of infections in infancy. Br J Nutr. 2011 Feb;105(3):409-16. doi: 10.1017/S0007114510003685. Epub 2010 Sep 24. PMID 20863419
- [Background] Luoto R, Ruuskanen O, Waris M, Kalliomaki M, Salminen S, Isolauri E. Prebiotic and probiotic supplementation prevents rhinovirus infections in preterm infants: a randomized, placebo-controlled trial. J Allergy Clin Immunol. 2014 Feb;133(2):405-13. doi: 10.1016/j.jaci.2013.08.020. Epub 2013 Oct 13. PMID 24131826
- [Background] Giovannini M, Agostoni C, Riva E, Salvini F, Ruscitto A, Zuccotti GV, Radaelli G; Felicita Study Group. A randomized prospective double blind controlled trial on effects of long-term consumption of fermented milk containing Lactobacillus casei in pre-school children with allergic asthma and/or rhinitis. Pediatr Res. 2007 Aug;62(2):215-20. doi: 10.1203/PDR.0b013e3180a76d94. PMID 17597643
- [Background] Kukkonen K, Savilahti E, Haahtela T, Juntunen-Backman K, Korpela R, Poussa T, Tuure T, Kuitunen M. Long-term safety and impact on infection rates of postnatal probiotic and prebiotic (synbiotic) treatment: randomized, double-blind, placebo-controlled trial. Pediatrics. 2008 Jul;122(1):8-12. doi: 10.1542/peds.2007-1192. PMID 18595980
- [Background] Leyer GJ, Li S, Mubasher ME, Reifer C, Ouwehand AC. Probiotic effects on cold and influenza-like symptom incidence and duration in children. Pediatrics. 2009 Aug;124(2):e172-9. doi: 10.1542/peds.2008-2666. Epub 2009 Jul 27. PMID 19651563
- [Background] Rautava S, Salminen S, Isolauri E. Specific probiotics in reducing the risk of acute infections in infancy--a randomised, double-blind, placebo-controlled study. Br J Nutr. 2009 Jun;101(11):1722-6. doi: 10.1017/S0007114508116282. Epub 2008 Nov 6. PMID 18986600
- [Background] Rerksuppaphol S, Rerksuppaphol L. Randomized controlled trial of probiotics to reduce common cold in schoolchildren. Pediatr Int. 2012 Oct;54(5):682-7. doi: 10.1111/j.1442-200X.2012.03647.x. Epub 2012 Jul 10. PMID 22507276
- [Background] Sazawal S, Dhingra U, Hiremath G, Sarkar A, Dhingra P, Dutta A, Verma P, Menon VP, Black RE. Prebiotic and probiotic fortified milk in prevention of morbidities among children: community-based, randomized, double-blind, controlled trial. PLoS One. 2010 Aug 13;5(8):e12164. doi: 10.1371/journal.pone.0012164. PMID 20730056
- [Background] Weizman Z, Asli G, Alsheikh A. Effect of a probiotic infant formula on infections in child care centers: comparison of two probiotic agents. Pediatrics. 2005 Jan;115(1):5-9. doi: 10.1542/peds.2004-1815. PMID 15629974
- [Background] King S, Glanville J, Sanders ME, Fitzgerald A, Varley D. Effectiveness of probiotics on the duration of illness in healthy children and adults who develop common acute respiratory infectious conditions: a systematic review and meta-analysis. Br J Nutr. 2014 Jul 14;112(1):41-54. doi: 10.1017/S0007114514000075. Epub 2014 Apr 29. PMID 24780623
- [Background] Garcia Jimenez E, Cortes Rubio JA, Oliart Delgado de Torres S, Reig del Moral C, Herrera Martin M, Garcia Velazquez J, Cuadrado Bello P. [Systemic lupus erythematosus and pancreatitis. Apropos of a case]. An Esp Pediatr. 1992 Apr;36(4):311-3. No abstract available. Spanish. PMID 1605420
- [Background] Gleeson M, Bishop NC, Oliveira M, McCauley T, Tauler P, Lawrence C. Effects of a Lactobacillus salivarius probiotic intervention on infection, cold symptom duration and severity, and mucosal immunity in endurance athletes. Int J Sport Nutr Exerc Metab. 2012 Aug;22(4):235-42. doi: 10.1123/ijsnem.22.4.235. Epub 2012 May 10. PMID 22645171
- [Background] Pylkkanen K. Proceedings: Drug abuse as a symptom of negative identity crisis. Case report. Acta Paediatr Scand Suppl. 1975;(256):37. doi: 10.1111/j.1651-2227.1975.tb17595.x. No abstract available. PMID 1065193
- [Background] Rizzardini G, Eskesen D, Calder PC, Capetti A, Jespersen L, Clerici M. Evaluation of the immune benefits of two probiotic strains Bifidobacterium animalis ssp. lactis, BB-12(R) and Lactobacillus paracasei ssp. paracasei, L. casei 431(R) in an influenza vaccination model: a randomised, double-blind, placebo-controlled study. Br J Nutr. 2012 Mar;107(6):876-84. doi: 10.1017/S000711451100420X. Epub 2011 Sep 7. PMID 21899798
- [Background] de Vrese M, Winkler P, Rautenberg P, Harder T, Noah C, Laue C, Ott S, Hampe J, Schreiber S, Heller K, Schrezenmeir J. Probiotic bacteria reduced duration and severity but not the incidence of common cold episodes in a double blind, randomized, controlled trial. Vaccine. 2006 Nov 10;24(44-46):6670-4. doi: 10.1016/j.vaccine.2006.05.048. Epub 2006 Jun 6. PMID 16844267
- [Background] Ghadimi D, Folster-Holst R, de Vrese M, Winkler P, Heller KJ, Schrezenmeir J. Effects of probiotic bacteria and their genomic DNA on TH1/TH2-cytokine production by peripheral blood mononuclear cells (PBMCs) of healthy and allergic subjects. Immunobiology. 2008;213(8):677-92. doi: 10.1016/j.imbio.2008.02.001. Epub 2008 Apr 2. PMID 18950596
- [Background] Yasui H, Shida K, Matsuzaki T, Yokokura T. Immunomodulatory function of lactic acid bacteria. Antonie Van Leeuwenhoek. 1999 Jul-Nov;76(1-4):383-9. PMID 10532394
- [Background] Hori T, Kiyoshima J, Shida K, Yasui H. Effect of intranasal administration of Lactobacillus casei Shirota on influenza virus infection of upper respiratory tract in mice. Clin Diagn Lab Immunol. 2001 May;8(3):593-7. doi: 10.1128/CDLI.8.3.593-597.2001. PMID 11329464
- [Background] Stahl B, Barrangou R. Complete genome sequences of probiotic strains Bifidobacterium animalis subsp. lactis B420 and Bi-07. J Bacteriol. 2012 Aug;194(15):4131-2. doi: 10.1128/JB.00766-12. PMID 22815448
- [Background] Altermann E, Russell WM, Azcarate-Peril MA, Barrangou R, Buck BL, McAuliffe O, Souther N, Dobson A, Duong T, Callanan M, Lick S, Hamrick A, Cano R, Klaenhammer TR. Complete genome sequence of the probiotic lactic acid bacterium Lactobacillus acidophilus NCFM. Proc Natl Acad Sci U S A. 2005 Mar 15;102(11):3906-12. doi: 10.1073/pnas.0409188102. Epub 2005 Jan 25. PMID 15671160
- [Background] Hempel S, Newberry S, Ruelaz A, Wang Z, Miles JN, Suttorp MJ, Johnsen B, Shanman R, Slusser W, Fu N, Smith A, Roth B, Polak J, Motala A, Perry T, Shekelle PG. Safety of probiotics used to reduce risk and prevent or treat disease. Evid Rep Technol Assess (Full Rep). 2011 Apr;(200):1-645. PMID 23126627
- [Background] West NP, Horn PL, Pyne DB, Gebski VJ, Lahtinen SJ, Fricker PA, Cripps AW. Probiotic supplementation for respiratory and gastrointestinal illness symptoms in healthy physically active individuals. Clin Nutr. 2014 Aug;33(4):581-7. doi: 10.1016/j.clnu.2013.10.002. Epub 2013 Oct 10. PMID 24268677
- [Background] Jansen K, Blimkie D, Furlong J, Hajjar A, Rein-Weston A, Crabtree J, Reikie B, Wilson C, Kollmann T. Polychromatic flow cytometric high-throughput assay to analyze the innate immune response to Toll-like receptor stimulation. J Immunol Methods. 2008 Jul 31;336(2):183-92. doi: 10.1016/j.jim.2008.04.013. Epub 2008 May 16. PMID 18565537
- [Background] Corbett NP, Blimkie D, Ho KC, Cai B, Sutherland DP, Kallos A, Crabtree J, Rein-Weston A, Lavoie PM, Turvey SE, Hawkins NR, Self SG, Wilson CB, Hajjar AM, Fortuno ES 3rd, Kollmann TR. Ontogeny of Toll-like receptor mediated cytokine responses of human blood mononuclear cells. PLoS One. 2010 Nov 30;5(11):e15041. doi: 10.1371/journal.pone.0015041. PMID 21152080
- [Background] Blimkie D, Fortuno ES 3rd, Yan H, Cho P, Ho K, Turvey SE, Marchant A, Goriely S, Kollmann TR. Variables to be controlled in the assessment of blood innate immune responses to Toll-like receptor stimulation. J Immunol Methods. 2011 Mar 7;366(1-2):89-99. doi: 10.1016/j.jim.2011.01.009. Epub 2011 Jan 28. PMID 21277305
- [Background] Santos Rocha C, Gomes-Santos AC, Garcias Moreira T, de Azevedo M, Diniz Luerce T, Mariadassou M, Longaray Delamare AP, Langella P, Maguin E, Azevedo V, Caetano de Faria AM, Miyoshi A, van de Guchte M. Local and systemic immune mechanisms underlying the anti-colitis effects of the dairy bacterium Lactobacillus delbrueckii. PLoS One. 2014 Jan 21;9(1):e85923. doi: 10.1371/journal.pone.0085923. eCollection 2014. PMID 24465791
- [Background] de Roock S, van Elk M, van Dijk ME, Timmerman HM, Rijkers GT, Prakken BJ, Hoekstra MO, de Kleer IM. Lactic acid bacteria differ in their ability to induce functional regulatory T cells in humans. Clin Exp Allergy. 2010 Jan;40(1):103-10. doi: 10.1111/j.1365-2222.2009.03344.x. Epub 2009 Oct 7. PMID 19817754
- [Background] Singh AM, Dahlberg P, Burmeister K, Evans MD, Gangnon R, Roberg KA, Tisler C, Dasilva D, Pappas T, Salazar L, Lemanske RF Jr, Gern JE, Seroogy CM. Inhaled corticosteroid use is associated with increased circulating T regulatory cells in children with asthma. Clin Mol Allergy. 2013 Jan 25;11(1):1. doi: 10.1186/1476-7961-11-1. PMID 23347774
- [Background] Nettenstrom L, Alderson K, Raschke EE, Evans MD, Sondel PM, Olek S, Seroogy CM. An optimized multi-parameter flow cytometry protocol for human T regulatory cell analysis on fresh and viably frozen cells, correlation with epigenetic analysis, and comparison of cord and adult blood. J Immunol Methods. 2013 Jan 31;387(1-2):81-8. doi: 10.1016/j.jim.2012.09.014. Epub 2012 Oct 9. PMID 23058673

DOCUMENTS (1):
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT02687503/Prot_000.pdf